CLINICAL TRIAL: NCT05249712
Title: Medical Ethics Committee of Nanjing Drum Tower Hospital Affiliated to Medical School of Nanjing University
Brief Title: Efficacy and Safety of Darolutamide Combined With ADT in High-risk/Very High-risk Localized Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Collaborators: First Affiliated Hospital of Zhejiang University (Other); The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Hongqian Guo, Chief physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IUNU-PC-112
Record Dates: First submitted 2022-02-10; First posted 2022-02-22 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — darolutamide; Androgen Antagonists

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ADT with Darolutamide (Experimental): Pathological response rate after radical prostatectomy with dalotamide combined with androgen deprivation therapy (ADT) in neoadjuvant therapy for surgically resectable high-risk or very high-risk prostate cancer.
  Duration of treatment: 28-day cycle of darotamide treatment and 6 cycles of neoadjuvant therapy. ADT treatment continued during neoadjuvant therapy and was discontinued after surgery.
  Adjusted dosing: When the serum testosterone concentration cannot be maintained at <50 ng/dL, the dose and type of ADT can be adjusted. Investigators can adjust the dose of darostatide according to the situation.
  Interventions: Drug: Darolutamide 300 mg; Other: Androgen deprivation therapy

INTERVENTIONS:
Drug: Darolutamide 300 mg — 600 mg (300 mg × 2 tablets) twice daily with meals, equivalent to a total daily dose of 1200 mg.
  Other Names: Nubeqa, BAY1841788
Other: Androgen deprivation therapy — The ADT regimen used by each patient will be determined by the investigator, and the dose and frequency of administration will be consistent with the prescribing information.
  Other Names: ADT

SUMMARY:
This trial aims to evaluate the efficacy and safety of neoadjuvant therapy with Darolutamide combined with Androgen-Deprivation Therapy in High-risk/Very high-risk localized prostate cancer. This trial is A prospective, single-arm, multicenter clinical trial. Treatment cycle is 24 weeks,

DETAILED DESCRIPTION:
High risk prostate cancer (PCa) had worse outcomes on radical treatment results, short-time oncological results, even cancer-specific survival, than those low or mediate risk PCa. Neoadjuvant treatment before radical prostatectomy had been proven to get some benefits on peri-operation results, especially on reduction of tumor volume and minimization of biochemical recurrence. This study will evaluate the efficacy and safety of androgen deprivation therapy (ADT) with Darolutamide in neoadjuvant therapy for surgically resectable high-risk or very high-risk PCa.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be ≥ 18 and ≤75 years of age；
2. All patients must have a histologically or cytologically diagnosis of prostate cancer，without distant metastasis, and suitable for radical prostatectomy；
3. All patients meet at least one of the following criteria：

   1. multi-parameter MRI or PSMA PET / CT shows clinical staging of primary tumor ≥ T3；
   2. Gleason score of primary tumor ≥ 8；
   3. prostate specific antigen (PSA) ≥20 ng/ml； d) Radiographic assessment of regional lymph node metastases (N1)；
4. Eastern Cooperative Oncology Group (ECOG) physical condition score 0- 1；
5. Patients must have adequate organ function： hematologic function：within 28 days prior to registration as evidenced by: white blood cell (WBC) ≥ 4.0 × 109 / L, platelets≥ 100 × 109 / L, hemoglobin ≥ 9 g / dL and international normalized ratio (INR) < 1.5； renal function：within 28 days prior to registration, as evidenced by serum creatinine ≤2×ULN； hepatic function: within 28 days prior to registration, as evidenced by: total bilirubin (TBIL)≤1.5 x upper limit of normal (ULN),and SGOT (AST) and SGPT (ALT) ≤ 2.5 x ULN；
6. Patients must participate voluntarily and sign an informed consent form (ICF), indicating that they understand the purpose and required procedures of the study, and are willing to participate in. Patients must be willing to obey the prohibitions and restrictions specified in the research protocol.
7. Patients of childbearing potential must be willing to take high-efficiency contraceptive measures during the study period and within 120 days after the last dose of treatment.

Exclusion Criteria:

1. Patients with prostate having neuroendocrine, small cell, or sarcoma-like features are not eligible.
2. Patients with low-risk and medium-risk, localized prostate cancer (the following conditions are met at the same time) are not eligible: multiparameter MRI or PSMA PET / CT shows clinical staging of primary tumor < T3, Gleason score of primary tumor < 8, and prostate specific antigen (PSA)。
3. Patients with clinical or radiological evidence of regional or extra-regional lymph node metastases or bone metastases or visceral metastases are not eligible.（any M1）。
4. Patients who have previously received androgen deprivation therapy (medical or surgical) more than 3 months or focal treatment of prostate cancer or prostate cancer radiotherapy or prostate cancer chemotherapy are not eligible
5. Patients with severe or uncontrolled concurrent infections are not eligible。
6. Patients must not have New York Heart Association Class III or IV congestive heart failure at the time of screening. Patients must not have any thromboembolic event, unstable angina pectoris, myocardial infarction within 6 months prior to registration.
7. Patients must not have uncontrolled severe hypertension, persistent uncontrolled diabetes, oxygen-dependent lung disease, chronic liver disease, or HIV infection.
8. Patients must not have had other malignancies other than prostate cancer in the past 5 years, but cured basal cell or squamous cell skin cancers can be enrolled.
9. The patient is mentally ill, mentally disabled or incapable of giving informed consent

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Pathological Response Rate （pCR or MRD） | up to 8months
  Pathological Response Rate is defined as the pCR(Pathologic Complete Response Rate) or MRD (Proportion of Subjects With Minimal Residual Disease) Pathologic Complete Response Rate is defined as the proportion of subjects with no morphologically recognizable cancer cell in tumor specimens after radical prostatectomy.
  Proportion of Subjects With Minimal Residual Disease is defined as the proportion of subjects that have residual tumors with maximum diameter of 5 mm or less after radical prostatectomy or residual cancer burden <0.25cm3.

SECONDARY OUTCOMES:
AEs/SAEs | Baseline up to 30 days after the last dose of study drug or before initiation of a new antitumor treatment, whichever occurred first
  The level of AEs defined by NCI-CTCAE v5.0. Safety assessments will be assessed and documented after initiation of study drug, regardless of relationship to study drug.
  The level of complications defined by Clavien-Dindo classification.
PSA biochemical progression-free survival rate | 3 years
  Defined as the proportion of patients who did not experience biochemical progression or death within 3 years of initiation of darotamide treatment; biochemical progression was defined as an increase in serum PSA level to >0.2 ng/ml with 2 consecutive increases at least 3 months apart
Rate of Positive Surgical Margins | up to 8 months
  The proportion of subjects with positive surgical margins after radical prostatectomy
Rate of Stage Degradation | up to 8 months
  The proportion of subjects whose tumor clinical or pathological stage degradation after neoadjuvant therapy.
PSA response rate | up to 2 years
  The proportion of subjects with a ≥98% reduction in nadir PSA from baseline PSA during neoadjuvant therapy

OTHER OUTCOMES:
Change From Baseline in Quality of Life as assessed by FACT-P | up to 2 years
  Defined by Functional Assessment of Cancer Therapy-Prostate (FACT-P) questionnaire
Change From Baseline in Quality of life as assessed by BPI-SF | up to 2 years
  Defined by worst pain item based on BPI-SF questionnaire.
Change From Baseline in Quality of life as assessed by EPIC-26 | up to 2 years
  Defined by EPIC-26 questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Hongqian Guo, Phd, Principal Investigator — Nanjing Drum Tower Hospital, affiliated to medical school of Nanjing University
Locations (1):
- Hongqian Guo, Nanning, Jiangsu, China

REFERENCES:
- [Derived] Zhang X, Zhou F, Lu T, Zhang S, Wei X, Qiu X, Xu L, Guo H, Zhuang J. Neoadjuvant darolutamide plus androgen deprivation therapy for high-risk and locally advanced prostate cancer: a multicenter, open-label, single-arm, phase II trial. World J Urol. 2025 Jan 3;43(1):58. doi: 10.1007/s00345-024-05412-4. PMID 39751962